CLINICAL TRIAL: NCT02955173
Title: Significance of Circulating Tumor Cells (CTC) Detected by the CTCBIOPSY System as Potential Blood-based Biomarkers in Providing Prognostic and Predictive Information for Surgical Treatment of Gastric and Rectal Cancer
Brief Title: Significance of Circulating Tumor Cells in the Treatment of Gastric and Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Sanyuan Hu, Dr.& Prof., Qilu Hospital of Shandong University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2016YFC0106003
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Circulating Tumor Cells; Colorectal Cancer; Gastric Cancer
MeSH Terms: conditions — Neoplastic Cells, Circulating; Colorectal Neoplasms; Stomach Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Open surgery of rectal cancer (Experimental): Patients undergoing rectal cancer resection in an open approach
  Interventions: Procedure: Surgery
- Laparoscopic surgery of rectal cancer (Experimental): Patients undergoing rectal cancer resection in a laparoscopic approach
  Interventions: Procedure: Surgery
- Open surgery of gastric cancer (Experimental): Patients undergoing gastric cancer resection in an open approach
  Interventions: Procedure: Surgery
- Laparoscopic surgery of gastric cancer (Experimental): Patients undergoing gastric cancer resection in a laparoscopic approach
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Laparoscopic or open surgery for resection of gastric or rectal cancer

SUMMARY:
The primary purpose of this study is to compare both short-term and long-term treatment effect of laparoscopic vs. open approach on progressive gastric and rectal cancer, based on circulating tumor cell (CTC) test results as well as disease-free survivals, and figure out principles of laparoscopic approach for progressive gastric and rectal cancer. Secondary purpose is to establish an evaluation system for laparoscopic surgery for progressive gastric and rectal cancer treatment using CTC as a biomarker.

DETAILED DESCRIPTION:
Laparoscopic surgery represents a milestone for treatment of gastric and rectal cancer, with advantages of minimal invasion and rapid recovery compared to open approach. However, for progressive gastric and rectal cancer, laparoscopic approach has not been officially promoted by NCCN guideline (2015).

Over the past decade, circulating tumor cells (CTCs), originated from a tumor cell, have been identified as potential blood-based biomarkers capable of providing prognostic and predictive Information.

In the present study, the investigators utilize the CTCBIOPSY® system (YZYBIO Company, Wuhan, China), which has been approved by CFDA (Chinese Food and Drug Administration), to detect CTCs, and try to compare both short-term and long-term treatment effect of laparoscopic vs. open approach on progressive gastric and rectal cancer, based on circulating tumor cell (CTC) test results as well as disease-free survivals, and figure out principles of laparoscopic approach for progressive gastric and rectal cancer. Secondary purpose is to establish an evaluation system for laparoscopic surgery for progressive gastric and rectal cancer treatment using CTC as a biomarker.

ELIGIBILITY:
Gastric cancer

Inclusion Criteria:

* Gastric cancer of stage II/III

Exclusion Criteria:

* History of malignant tumors
* Gastric cancer of stage Ⅳ
* Preoperative neoadjuvant chemotherapy
* History of upper abdominal surgery
* Severe other contradictions of surgery

Rectal cancer

Inclusion Criteria:

* Primary rectal carcinoma
* Single lesion
* No metastasis
* Sphincter-saving surgery available

Exclusion Criteria:

* History of malignant tumors
* Acute bowel obstruction, bleeding or perforation
* Tumor over 6cm in diameter or in severe adhesion with surrounded tissues
* Severe other contradictions of surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2016-12; Primary Completion 2020-12-14 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | Two years

SECONDARY OUTCOMES:
Circulating tumor cell (CTC) test | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Sanyuan Hu, M.D. Ph.D., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benson AB 3rd, Venook AP, Bekaii-Saab T, Chan E, Chen YJ, Cooper HS, Engstrom PF, Enzinger PC, Fenton MJ, Fuchs CS, Grem JL, Grothey A, Hochster HS, Hunt S, Kamel A, Kirilcuk N, Leong LA, Lin E, Messersmith WA, Mulcahy MF, Murphy JD, Nurkin S, Rohren E, Ryan DP, Saltz L, Sharma S, Shibata D, Skibber JM, Sofocleous CT, Stoffel EM, Stotsky-Himelfarb E, Willett CG, Gregory KM, Freedman-Cass D. Rectal Cancer, Version 2.2015. J Natl Compr Canc Netw. 2015 Jun;13(6):719-28; quiz 728. doi: 10.6004/jnccn.2015.0087. PMID 26085388
- [Background] Lowes LE, Bratman SV, Dittamore R, Done S, Kelley SO, Mai S, Morin RD, Wyatt AW, Allan AL. Circulating Tumor Cells (CTC) and Cell-Free DNA (cfDNA) Workshop 2016: Scientific Opportunities and Logistics for Cancer Clinical Trial Incorporation. Int J Mol Sci. 2016 Sep 8;17(9):1505. doi: 10.3390/ijms17091505. PMID 27618023